CLINICAL TRIAL: NCT04524572
Title: The Role of a Motion Sensor With Accompanying Web Application on Step Counts, Energy Balance, and Metabolic Markers in Nurses
Acronym: WALK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Jennifer Reed, Scientist, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20130429
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Cardiovascular Risk Factor; Cardiovascular Diseases
Keywords: cardiovascular disease; motor activity; woman; workplace; Delivery of health care
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individual Challenge (Experimental): Participants will be able to log onto their Tractivity® Online web account at any time during the 4-week intervention phase to track their daily step counts and physical activity expenditure
  Interventions: Behavioral: Motion sensor
- friend challenge (Experimental): Participants will be able to log onto their Tractivity® Online web account at any time during the 4-week intervention phase to track their daily step counts and physical activity expenditure in comparison to the group average of all participants randomized to the friend challenge.
  Interventions: Behavioral: Motion sensor
- Team challenge (Experimental): participants will be able to log onto their Tractivity® Online web account at any time during the 4-week intervention phase to track their teams' daily step counts and physical activity expenditure in comparison to the group average of other teams.
  Interventions: Behavioral: Motion sensor

INTERVENTIONS:
Behavioral: Motion sensor — To explore the role of a motion sensor with accompanying web application on step counts, energy balance, and metabolic markers in nurses

SUMMARY:
The purpose of this prospective randomized controlled trial is to explore the role of a motion sensor with accompany web application on step counts, energy balance, and metabolic markers in nurses. Additionally, eating behaviours, behavioural regulation in exercise, and mood states that may impact these parameters will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* 1. Participant must be a registered nurse with the University of Ottawa Heart Institute;

  2. Participant must be 18 years of age or older;

  3. Participant must be able to walk unassisted;

  4. Participant is able and willing to provide informed consent.

Exclusion Criteria:

1. Participant is pregnant, lactating or planning to become pregnant during the study period;
2. Participant is unable to read and understand English;
3. Medical contraindications to exercise;
4. Already using a motion sensor device to track physical activity. -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-11-26 (Actual); Primary Completion 2014-04-25 (Actual); Study Completion 2015-08-01 (Actual)

PRIMARY OUTCOMES:
Step counts | 6 weeks during observation and 6 weeks during intervention
  All participants will be asked to wear a Tractivity® motion sensor device on their ankle for to assess their daily step count and physical activity energy expenditure

SECONDARY OUTCOMES:
Body Mass (kg) | Screening (week 1), Observation (weeks 2-5), during the intervention (weeks 6-9), post study at week 26 and week 52
  Body weight will be measured using a digital scale to the nearest 0.1 kilogram
Waist Circumference | Screening (week 1), Observation (weeks 2-5), during the intervention (weeks 6-9), post study at week 26 and week 52
  Waist circumference will be measured using a tape measure
Fat mass | Screening (week 1), Observation (weeks 2-5), during the intervention (weeks 6-9), post study at week 26 and week 52
  Fat mass will be measured using bioelectrical impedance analysis

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Brunet J, Black M, Tulloch HE, Pipe AL, Reid RD, Reed JL. Work-related factors predict changes in physical activity among nurses participating in a web-based worksite intervention: A randomized controlled trial. BMC Nurs. 2021 Nov 9;20(1):224. doi: 10.1186/s12912-021-00739-4. PMID 34749710
- [Derived] Brunet J, Tulloch HE, Wolfe Phillips E, Reid RD, Pipe AL, Reed JL. Motivation Predicts Change in Nurses' Physical Activity Levels During a Web-Based Worksite Intervention: Results From a Randomized Trial. J Med Internet Res. 2020 Sep 11;22(9):e11543. doi: 10.2196/11543. PMID 32915158